CLINICAL TRIAL: NCT02338258
Title: The Prospective、Randomized、Comparative Clinical Study About the Two Operation Methods Between Anti-rotational Plate Group and Exchanged Intramedullary Nailgroup to Treat the Nonunion of Long Tubular Bone After Intramedullary Nail Fixation
Brief Title: The Study of the Nonunion of Long Tubular Bone
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, Xianzhi Ma, Beijing Jishuitan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Z141107002514086
Record Dates: First submitted 2014-12-26; First posted 2015-01-14 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Diaphyses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The Anti-rotational plate group (Experimental): The method was used to control the rotational unstabilization at the fracture site
  Interventions: Device: Anti-rotational plate; Device: Exchanged Intramedullary nailing
- Exchanged Intramedullary nailing group (Placebo Comparator): the method Provided the axial and rotational stability
  Interventions: Device: Exchanged Intramedullary nailing

INTERVENTIONS:
Device: Anti-rotational plate
  Arms: The Anti-rotational plate group
Device: Exchanged Intramedullary nailing

SUMMARY:
The purpose of the study to supplied the diagnostic and treatment criteria of the nonunion of the long tubular bone after treatment of Intramedallery nailing

ELIGIBILITY:
Inclusion Criteria:

1. The patient who had the nonunion of long tubular bone
2. The patient who was the age of 14 ~ 65 years old.
3. The patient who complete the follow-up conditions.
4. The patient who has independent behavior ability.
5. The patient who volunteered for signed informed consent

Exclusion Criteria:

1. Infectious nonunion of the long turubar bone
2. Pathological fracture.
3. The immune system disease.
4. Cancer

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-09 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
The healing rate | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Bosong Zhang, MD, Principal Investigator — Jishuitan hospital in Beijing
Locations (1):
- The orthopaedic Trauma center of Jishuitan Hospital in Beijing, Beijing, Beijing Municipality, China